CLINICAL TRIAL: NCT00895232
Title: Iron Sucrose In The Treatment of Restless Legs Syndrome (RLS): The Safety of Three Dose Regimens as Evaluated by Clinical Assessments
Brief Title: Iron Sucrose In The Treatment of Restless Legs Syndrome: Safety of Three Dose Regimens as Evaluated by Clinical Assessments
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1VEN03032
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Results first posted 2015-06-10 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort I (Experimental): 500 mg dose Venofer over 4 hours
  Interventions: Drug: Cohort I
- Cohort II (Experimental): 500 mg Venofer infusion over 4-6 hours on Day 0 and repeated on Day 2 to 7
  Interventions: Drug: Cohort II
- Cohort III (Experimental): 500 mg Venofer over 6 hours, followed within 24 hours by 500 mg Venofer over 6 hours
  Interventions: Drug: Cohort III

INTERVENTIONS:
Drug: Cohort I
  Other Names: iron sucrose injection - Venofer
  Arms: Cohort I
Drug: Cohort II
  Other Names: iron sucrose injection - Venofer
  Arms: Cohort II
Drug: Cohort III
  Other Names: iron sucrose injection - Venofer
  Arms: Cohort III

SUMMARY:
Non-randomized open label Phase II clinical trial in which subjects meeting criteria for RLS were assigned to 1 of 3 treatment cohorts. The first cohort received one 500 mg IV iron sucrose infusion in 500 mL normal sterile saline (NSS) administered over four hours. The second cohort received two 500 mg IV iron sucrose infusions in 500mL of NSS administered over four to six hours on two separate dates, separated by two to seven days. The third cohort received two 500 mg IV iron sucrose infusions in at least 500 mL of NSS over six hours within 30 hours of the start of the first infusion. Cohorts were enrolled and treated subsequently.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent.
* Male or female subjects > 18 yrs. old.
* RLS signs and symptoms affirming diagnosis.
* A baseline score > or = to 15 is required on the International RLS Study Group Rating Scale (IRLSSG).
* At least one leg with an average baseline Periodic Leg Movement (PLM) while asleep > or = to 15 movements per hour by actigraphy.
* Subjects on dopa-adrenergic therapy or other RLS treatments must be off therapy at least one week before any baseline RLS assessments and actigraphy measurement are obtained.
* Subject has regular sleep hours between 9 p.m. and 9 a.m.
* Subjects at risk for pregnancy must have a negative pregnancy test at baseline and be practicing an acceptable form of birth control.

Exclusion Criteria:

* Known intolerance to Venofer.
* RLS which is ascribed to renal disease.
* RLS 2° to other CNS disease or injury.
* Any pain related or sleep related disorders which may confound the outcome measures.
* History of neuroleptic akinesia.
* Concurrent use of oral iron supplement.
* Parenteral iron use within the past 6 months.
* Active infection.
* Currently being treated for asthma.
* Severe peripheral vascular disease with significant skin changes.
* Seizure disorder currently being treated with medication.
* Serum ferritin level > 300 ng/mL or a TSAT > or = to 45% at baseline or a history of hemochromatosis.
* Significant cardiovascular or hepatic disease or any other pre-existing medical condition or disease which in the view of the investigator participation in this study would put the subject's disease management at risk or the subject would be unable to comply with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2003-11; Primary Completion 2005-08 (Actual); Study Completion 2005-11 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: November 14, 2003 - August 8, 2005 Locations: Hospitals and Medical Clinics
Pre-assignment Details: A Baseline score > or = to 15 was required on the International RLS Study Group (IRLSSG) Rating Scale. At least 1 leg was required to have an average baseline Periodic Leg Movement (PLM) while asleep > or = to 15 movements per hour by actigraphy.
Groups:
- Cohort I (Venofer 500mg x 1 Dose): Single 500 mg infusion of Venofer over 4 hours.
- Cohort II (Venofer 500mg X 2 Doses): A 500 mg infusion of Venofer over 4 to 6 hours on Day 0; with a second 500 mg infusion administered between Day 2 and Day 7.
- Cohort III (Venofer 500mg x 2 Doses): A 500 mg infusion of Venofer over 6 hours on Day 0, followed within 24 hours by a second 500 mg infusion of Venofer over 6 hours.
Period: Overall Study
Arm/Group | Cohort I (Venofer 500mg x 1 Dose) | Cohort II (Venofer 500mg X 2 Doses) | Cohort III (Venofer 500mg x 2 Doses)
Started | 7 | 6 | 8
Completed | 4 | 2 | 3
Not Completed | 3 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I (Venofer 500mg x 1 Dose) | Cohort II (Venofer 500mg X 2 Doses) | Cohort III (Venofer 500mg x 2 Doses) | Total
Number analyzed (Participants) | 7 | 6 | 8 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 8 | 18
  >=65 years | 2 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 11
  Male | 3 | 2 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Day 84 for International Restless Leg Syndrome Study Group (IRLSSG) Scale
Description: Validated rating scale of RLS symptoms (Range 1 [mild] - 40 [severe])
Time Frame: Baseline to Day 84
Population: Only subjects who completed the IRLSSG Rating Scale at baseline AND on Day 84.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cohort I (Venofer 500mg x 1 Dose) | Cohort II (Venofer 500mg X 2 Doses) | Cohort III (Venofer 500mg x 2 Doses)
Number analyzed (Participants) | 5 | 3 | 2
units on a scale | -2.4 (5.41) | -14.3 (5.03) | -16.0 (8.49)

2. Post Hoc Outcome: Percentage (%) of Subjects Responding to Treatment From Baseline to Day 84 Based on Global Assessments by the Examiner.
Description: Response is defined as any effect based on a scale of 0 through 4 where 0 = no effect, 1 = mild effect, 2 = moderate effect, 3 = marked effect, and 4 = dramatic effect.
Time Frame: Baseline to Day 84
Population: Only subjects who were evaluated at Baseline AND on Day 84
Measure: Number; unit: percent of participants
Arm/Group | Cohort I (Venofer 500mg x 1 Dose) | Cohort II (Venofer 500mg X 2 Doses) | Cohort III (Venofer 500mg x 2 Doses)
Number analyzed (Participants) | 7 | 3 | 3
percent of participants | 28.6 | 66.7 | 66.7

3. Secondary Outcome: Mean Change From Baseline to Day 84 for Total Periodic Limb Movements (PLM's)
Description: Quantifies amount of leg movement
Time Frame: Baseline to Day 84
Population: Only subjects who recorded PLM's/Hour at Baseline AND on Day 84.
Measure: Mean (Standard Deviation); unit: PLM's per hour
Arm/Group | Cohort I (Venofer 500mg x 1 Dose) | Cohort II (Venofer 500mg X 2 Doses) | Cohort III (Venofer 500mg x 2 Doses)
Number analyzed (Participants) | 3 | 2 | 1
PLM's per hour | -7.2 (24.12) | -75.0 (49.71) | -96.2 (0)

ADVERSE EVENTS:
Time Frame: 1 year and 9 months
Arm/Group | Cohort I (Venofer 500mg x 1 Dose) | Cohort II (Venofer 500mg X 2 Doses) | Cohort III (Venofer 500mg x 2 Doses)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6 | 1/8
Other Adverse Events (participants affected / at risk) | 5/7 | 4/6 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (Venofer 500mg x 1 Dose) (N=7) | Cohort II (Venofer 500mg X 2 Doses) (N=6) | Cohort III (Venofer 500mg x 2 Doses) (N=8)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort I (Venofer 500mg x 1 Dose) (N=7) | Cohort II (Venofer 500mg X 2 Doses) (N=6) | Cohort III (Venofer 500mg x 2 Doses) (N=8)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea NOS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension NOS (Vascular disorders) | 0 (0) | 3 (3) | 2 (2)
Injection site reaction NOS (General disorders) | 0 (0) | 1 (1) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Oedema NOS (General disorders) | 1 (1) | 2 (3) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 2 (2) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Phlebitis NOS (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic NOS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sweating increased (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria NOS (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Vomiting NOS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less